CLINICAL TRIAL: NCT03478137
Title: Effect of Continuous Positive Airway Pressure (CPAP) Treatment on Cognitive Ability in HIV+ Individuals With Obstructive Sleep Apnea (OSA): A Pilot Study
Brief Title: Obstructive Sleep Apnea, CPAP Treatment & Cognitive Ability in HIV
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: McGill University (Other)
Collaborators: VitalAire (Industry); ResMed (Industry)
Responsible Party: Principal Investigator, Marie-Josée Brouillette, Associate professor, McGill University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-3222
Record Dates: First submitted 2017-09-13; First posted 2018-03-27 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Hiv; Obstructive Sleep Apnea; Cognitive Change
Keywords: Cognition; Intervention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CPAP intervention (Experimental): Over the course of 4-7 months, participants will have to wear the CPAP every night, at least 4 hours per night.
  Interventions: Behavioral: CPAP intervention
- Control 1 (No Intervention): Eligible participants who declined to participate in the study. Their main study visit data will be used to compare with the intervention group.
- Control 2 (No Intervention): Eligible participants who were not approached, hence not given the opportunity to accept or decline. Their main study visit data will be used to compare with the intervention group.

INTERVENTIONS:
Behavioral: CPAP intervention — Participants who agree to participate will be evaluated by a sleep specialist who will confirm eligibility for CPAP treatment.Eligible participants will be referred to VitalAire for initiation of treatment following a standard protocol for CPAP use at home. CPAP treatment will continue until the next visit for the main study, between 4-7 months, based on the timing of the evaluations, after which the study will end.
  Arms: CPAP intervention

SUMMARY:
Obstructive sleep apnea (OSA) is a breathing disorder that is characterized by episodes of complete or partial cessation of respiration during sleep, associated with upper airway collapse, oxygen desaturation and sleep fragmentation. OSA is a condition frequently implicated in cognitive disturbances, as well as associated with health conditions such as hypertension, metabolic disturbances and heightened risk of heart disease, stroke and mortality. These conditions are also increased in persons living with HIV. Individuals suffering from OSA report an increase in daytime sleepiness, mood changes and decline in quality of life.OSA also portends economic and societal impact through lost productivity at work and motor vehicle accidents. The presence of OSA is therefore important to detect in those living with HIV as it is potentially treatable contributors to cognitive disturbances in HIV. Continuous Positive Airway Pressure (CPAP) is the recommended treatment of choice for OSA. CPAP has established efficacy in improving cognition (executive function, long-term verbal and visual memory, attention/vigilance and global cognitive functioning). Although CPAP has been associated with improvements in cognitive functioning in the general population, its effectiveness in improving cognition in HIV+ individuals has never been previously tested. Given that cognitive disturbances in this population are multi-factorial, determining whether treatment of OSA in this population improves cognition is key in improving the clinical management of HIV+ individuals, both for its negative impact on cognition, but also more generally for their health.

DETAILED DESCRIPTION:
Definition of obstructive sleep apnea:

Obstructive sleep apnea (OSA) is a breathing disorder that is characterized by episodes of complete or partial cessation of respiration during sleep, associated with upper airway collapse, oxygen desaturation and sleep fragmentation. The index commonly used to assess sleep disordered breathing (SDB) is the respiratory disturbance index (RDI), defined as the average number of respiratory disturbances (obstructive apneas, hypopneas, and respiratory event-related arousals [RERAs]) per hour. According to the Centers for Medicare & Medicaid Services criteria for the positive diagnosis and treatment of obstructive sleep apnea, a positive test for OSA is established if the RDI ≥ 15 events per hour.

Obstructive sleep apnea and cognition:

Obstructive sleep apnea (OSA) is a condition frequently implicated in cognitive disturbances. These cognitive deficits are common : for example, in a meta-analysis of individuals with OSA, information processing speed was reduced in as many as 75% of individuals compared with norm-referenced data. In addition to its negative impact on cognition, OSA is associated with health conditions such as hypertension, metabolic disturbances (including impaired glucose tolerance, insulin resistance and dyslipidemia) and heightening risk of heart disease, stroke and mortality, conditions also increased in persons living with HIV. Individuals suffering from OSA report an increase in daytime sleepiness, mood changes and decline in quality of life. OSA also portends economic and societal impact through lost productivity at work and motor vehicle accidents.The presence of OSA is therefore important to detect in those living with HIV as it is a potentially treatable contributors to cognitive disturbances in HIV.

Obstructive sleep apnea and HIV:

General population estimates of moderate to severe sleep-disordered breathing depend on criteria used and vary widely, from 6-13% of individuals, to up to 23% of women and 50% of men using modern criteria. This prevalence is increased in the HIV population. Based on data from the Multicenter AIDS Cohort Study (MACS, N=1896) and Women's Interagency HIV Study (WIHS, N=1976), HIV-infected individuals are more likely to be diagnosed with OSA than HIV-uninfected individuals when confounders such as age and body mass index were accounted for (Prevalence Ratio (PR) 1.42; p=0.01 and PR 2.10; p=0.002, respectively). HIV-infected individuals have many risk factors for OSA including a high rate of obesity: >60% of HIV-infected women in the WIHS and >40% of HIV-infected men and MACS.

Traditional risk factors associated with OSA include advanced age, male gender, large neck circumference, obesity and hypertension. However, these traditional clinical indicators of OSA may be less salient in the presence of HIV infection. In a large observational study, those with HIV and OSA were more likely to be younger, have lower body-mass-indexes and were less likely to have hypertension than those without HIV infection. As a result of this different risk profile, the presence of OSA in HIV+ individuals was more often undiagnosed, underscoring the need for a higher index of suspicion in the presence of HIV infection.

Treatment of obstructive sleep apnea and its impact on cognition:

Continuous Positive Airway Pressure (CPAP) is the recommended treatment of choice for OSA. A CPAP device includes a pump which delivers air via a mask covering the nose or mouth while a person in sleeping. The flow of air generates positive pressure, which opens the airways, preventing soft tissue collapse.

CPAP has established efficacy in improving cognition. A meta-review involving review articles meeting pre-determined strict criteria, concluded that CPAP use improved executive function, long-term verbal and visual memory, attention/vigilance and global cognitive functioning. Another meta-analysis also found that individuals with OSA demonstrated medium to very large impairments executive dysfunction, independent of age and disease severity, which showed small to moderate improvements following CPAP treatment. In the context of Alzheimer's disease, Ancoli-Israel et al. conducted a randomized double-blind placebo-controlled trial to determine whether CPAP use resulted in improvements in neuropsychological test scores. Although the study was underpowered to make definitive conclusions about improvements within specific cognitive constructs, exploratory post hoc examination of score changes suggested that CPAP use by individuals with OSA yielded some benefits; these included improvements in episodic verbal learning and memory and some aspects of executive functioning such as cognitive flexibility and mental processing speed.

Although CPAP has been associated with improvements in cognitive functioning in the general population, its effectiveness in improving cognition in HIV+ individuals has never been previously tested. Given that the cognitive disturbances in this population are multi-factorial, determining whether treatment of OSA in this population improves cognition is key in improving the clinical management of HIV+ individuals, both for its negative impact on cognition but also more generally for their health.

Obstructive sleep apnea in the cohort "Understanding and Optimizing Brain Health Now".

Cohort participants (N=840) are studied prospectively over a 27-month period with visits every 9 months. Patients complete a computer-based evaluation of cognitive ability, the B-CAM, as well as questionnaires on socio-demographic characteristics, symptom status, functional status, health perception and quality of life. Given the high prevalence of OSA reported in the population, participants complete questions that, combined with other values already documented, support the scoring of two screening questionnaires for OSA, the Berlin and the STOP-Bang. Selected cohort members at the Montreal sites who screen positive for the presence of OSA will be invited to participate in the study.

This study is part of a larger project based upon a cohort multiple randomized controlled design. Within a fully characterized cohort (N=840) which is followed over time, people meeting the specific criteria for one or more interventions (here CPAP) are identified and a sample is randomly selected to receive the intervention; the remaining eligible persons who do not receive the intervention serve as controls. This design, when operationalized for one intervention, yields three cohorts: (i) the intervention cohort comprising all those approached who agreed to enter; (ii) the refuser cohort comprising all those approached who declined entry; and (iii) control cohort comprising eligible persons who were not approached, and hence were not given the opportunity to accept or decline. For the CPAP intervention, the duration of the study is 4-7 months.

Eligible patients will be identified among the Montreal participants (N=500) in the "Understanding and Optimizing Brain Health Now" cohort study who have screened positive for the possible presence of sleep apnea on either the Berlin or the STOP-Bang and experience some cognitive difficulties as measured by the B-CAM (≤ 29).

Participants will undergo a polysomnography and will be evaluated by a sleep specialist who will confirm the presence of sleep apnea and eligibility for CPAP treatment. Eligible participants will be referred to VitalAire for initiation of treatment, following a standard protocol for use in the home. CPAP treatment will continue until the next visit for the main study, between 4-7 months based on the timing of the evaluations, after which the OSA study will end.

ELIGIBILITY:
Inclusion Criteria:

* Participants in the cohort study "Understanding and Optimizing Brain Health in HIV Now"
* Screened positive for OSA using the Berlin or the STOP-BANG (completed as part of the main study visits)
* Have been on a stable HAART regimen for > 6 months
* B-CAM ≤ 29
* Have not had a change in medications that could potentially interfere with sleep or cognition in the past 4 months.
* Willing to use CPAP as per instructions
* Able to comply with follow-up visit assessments
* Able to communicate in English or French
* Have at least one remaining visit in the main cohort study

Exclusion Criteria:

* Already treated for OSA
* Ongoing involvement in night shift work
* Presence of restless legs syndrome requiring immediate specific treatment

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2017-06-05 (Actual); Primary Completion 2021-09-13 (Estimated); Study Completion 2021-09-13 (Estimated)

PRIMARY OUTCOMES:
Changes in Cognitive Performance measure (B-CAM) | Up to 5 months before the beginning of the intervention and up to 1 month after the end of the intervention.
  The research team will be looking at changes on the B-CAM (brief cognitive ability measure) pre- and post-intervention

SECONDARY OUTCOMES:
Changes Self-reported cognitive difficulties (C3Q) | One week before the beginning of the intervention and up to 4 weeks after the end of the intervention
  The Communicating Cognitive Concerns Questionnaire evaluates cognitive concerns participants may have.
Adherence to the CPAP treatment | During the treatment (between 4 to 7 months)
  The CPAP device has a telemonitoring function. The data obtained yields a continuous metric of sleep-minutes of use

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Josée Brouillette, MD, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre; Lesley K Fellows, MD/DPhil, Principal Investigator — McGill University
Locations (1):
- McGill University Health Center, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-01-23): https://cdn.clinicaltrials.gov/large-docs/37/NCT03478137/Prot_000.pdf